CLINICAL TRIAL: NCT05323032
Title: Normal Multifocal Electroretinogram in Egyptian Population.
Brief Title: Multifocal Electroretinogram in Normal Egyptian Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC 5-22
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Retinal Disease; Healthy Population
Keywords: normal; electroretinogram; delta population
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Intervention Model Description: Multifocal electroretinogram in normal population
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal subjects (Experimental): Normal subjects at banha university that are seeking regular ophthalmic check-up.
  Interventions: Device: Multifocal electroretinogram (mf-ERG) by electroretinogram device

INTERVENTIONS:
Device: Multifocal electroretinogram (mf-ERG) by electroretinogram device — Measurement of mf-ERG parameters with 61 stimulus elements to asses amplitude of waves in nano volt/degree square (nv/deg2) and latency in millisecond (msec) as measured by electroretinogram device.

SUMMARY:
Studying normal subjects to create unique normal database for multifocal electroretinogram (mf-ERG) in specific population.

DETAILED DESCRIPTION:
Normal parameters for electroretinogram (ERG) is important in studying specific population, studying normal subjects is important to create specific normal database for each population. This will help in accurate differentiation for various ocular diseases and in research trials.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects seeking regular ophthalmic check-up at banha university hospital.

Exclusion Criteria:

* Any retinal diseases that may affects mf-ERG waves.
* Subjects with best corrected visual acuity less than 0.7 in decimal form at time of examination.
* Refractive errors more than 0.5 diopter as measured by autorefractometer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Amplitude of waves in nv/deg2 | immediately after mf-ERG diagnostic test for each eye.
  Measurement of the amplitude of N1 and P1 waves.
Latency of waves in msec. | immediately after mf-ERG diagnostic test for each eye.
  Measurement of the latency of N1 and P1 waves.

SECONDARY OUTCOMES:
Difference between different age groups in mf-ERG readings. | immediately after mf-ERG diagnostic test for each eye.
  Statistical analysis for mf-ERG amplitude and latency in different age groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Tabl, MD, Study Chair — Benha University
Locations (1):
- Ahmed Abdelshafy Tabl, Banhā, Banha, Egypt

IPD SHARING:
Plan to Share IPD: Undecided